CLINICAL TRIAL: NCT02230059
Title: Treatment Patterns in Metastatic Castration-Resistance Prostate Cancer (mCRPC): Real Life Analysis In Brazilian Oncology Centers (REALIST-PRO)
Brief Title: Study to Assess the Treatment Patterns in Metastatic Castration-Resistance Prostate Cancer (mCRPC)
Acronym: REALIST-PRO
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100943; 212082PCR0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; observational Study; Metastatic castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic Castration-resistant Prostate Cancer: Medical charts of participants with metastatic castration-resistant prostate cancer will be observed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Medical charts of participants with metastatic castration-resistant prostate cancer will be observed.

SUMMARY:
The purpose of this study is to assess the treatment patterns in participants with metastatic castration-resistant prostate cancer (mCRPC). Additionally, participant's demographic and clinical characteristics, skeletal-related events, criteria used to define CRPC, prostate specific antigen (PSA) levels and pain related to disease and overall survival will be observed.

DETAILED DESCRIPTION:
This is an observational (study in which participants identified as belonging to study groups are assessed for biomedical or health outcomes), longitudinal (correlational research study that involves repeated observations of the same variables over long periods of time) and retrospective (study looking back over past experience) study to describe the treatment patterns in mCRPC. Treatment patterns will be assessed by collecting medical charts from participants diagnosed with mCRPC in or prior 2009. Primarily, percentage of participants who received therapy as first line treatment will be assessed. All adverse events associated with the use of Sponsor drugs will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Report of previous surgical or medical castration
* Castration-resistant prostate cancer (CRPC) diagnosis in or before 2009
* Metastatic disease documented by positive bone scan or metastatic lesions on computed tomography or magnetic resonance imaging in or before 2009. If lymph node metastasis is the only evidence of metastasis, it must be 2 centimeters (cm) in diameter

Exclusion Criteria:

* Participation in any investigational drug or device study or early access programme

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male participants with history of prostatic cancer and metastatic castration-resistant prostate cancer (mCRPC) from Brazil will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Treated With Chemotherapy in First Line Therapy | Day 1
  Participants treated with chemotherapy in first line therapy will be reported.
Percentage of Participants Treated With Other Therapies in First Line Therapy | Day 1
  Participants treated with other therapies including secondary hormone therapy, steroids, radiation therapy, radionuclide therapy, bisphosphonates and best supportive care in first line therapy will be reported.
Percentage of Participants Treated With Chemotherapy in Second Line Therapy | Day 1
  Participants who were treated with chemotherapy in second line therapy will be reported.
Percentage of Participants Treated With Other Therapies in Second Line Therapy | Day 1
  Participants treated with other therapies including secondary hormone therapy, steroids, radiation therapy, radionuclide therapy, bisphosphonates and best supportive care in second line therapy will be reported.

SECONDARY OUTCOMES:
Eastern Cooperative Oncology Group (ECOG) Performance Status | Day 1
  ECOG performance status is a scale that measures how cancer affects the daily life of a participant on an ordinal scale from grade 0 (best) to grade 5 (worst).
Number of Participants with Comorbidities | Day 1
  Participants with comorbidities such as hypertension, diabetes, cardiac diseases, congestive cardiac failure, thyroid diseases and stroke will be reported.
Blood Prostate Specific Antigen (PSA) levels | Day 1
  Blood PSA levels will be reported.
Number of participants With Bone or Visceral Metastasis | Day 1
  Participants with bone or visceral metastasis will be reported.
Assessment of Pain Related With Disease | Day 1
  Pain will be assessed by reviewing the charts having information regarding pain (bone or other sites).
Number of Participants With Gleason score | Day 1
  Gleason scoring is used to grade tumors. A primary grade is assigned to the most common tumor pattern (how the cancer cells look under a microscope), and a second grade to the next most common pattern. The two grades are added together to get a GS. Gleason grade range= 1-5; 5=worst prognosis. GS range=2-10; 10=worst prognosis. Improvement is defined as a decrease in GS from a Baseline score of 6 (GS<=6; includes no cancer); worsening is defined as an increase in GS from a baseline score of 6 (GS >6).
Percentage of Participants With Skeletal Related Events (SREs) | Day 1
  SREs include vertebral collapse, bone fractures, spinal cord compression, bone surgery and radiotherapy for bone complications.
Number of Participants who were used to define mCRPC Criteria | Day 1
  Participants with criteria used to define mCRPC as described by European Association of Urology (EAU) International Guidelines will be reported.
Percentage of Participants Who Received Therapies After Second Line | Day 1
  Participants who received therapies after second line will be reported.
Overall Survival | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- Brazil (10):
  - Brasília
  - Curitiba
  - Distrito Federal
  - Florianópolis
  - Goiânia
  - Ijuí
  - Jaú
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo